CLINICAL TRIAL: NCT02262468
Title: Review of 750 36mm MOM Hip Replacements ( Pinnacle/Corail) With up to 6 Year Follow up
Brief Title: Warwick Metal On Metal Study
Status: Completed | Type: Observational
Sponsor: South Warwickshire NHS Foundation Trust (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Principal Investigator, Stephen Young, consultant orthopaedic surgeon, South Warwickshire NHS Foundation Trust
Other Study IDs: IIS2012012
Record Dates: First submitted 2014-10-07; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Metal Hip Replacement
Keywords: retrospective analysis
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MOM total hip replacements: all patients with MOM 36mm hip replacements
  Interventions: Radiation: x ray

INTERVENTIONS:
Radiation: x ray

SUMMARY:
assess results of metal on metal hip replacements carried out at warwick hospital

DETAILED DESCRIPTION:
Resurfacing and XL head hip replacements have not done as well as expected. The ASR implant has been withdrawn. Recent publications and media appearances by Tony Nargol, an orthopaedic surgeon, have suggested 36mm metal on metal replacements. I intend to report the results of this series.

ELIGIBILITY:
Inclusion Criteria:

* All patients with 36mm metal on metal hips

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with 36mm metal on metal hips
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Oxford hip score | 6 years